CLINICAL TRIAL: NCT03345940
Title: A Multicentric Randomized PRAGmatic Trial to Compare the Effectiveness of Fingolimod Versus Dimethyl-Fumarate on Patient Overall Disease Experience in Relapsing Remitting Multiple Sclerosis: Novel Data to Inform Decision-makers
Brief Title: Fingolimod Versus Dimethyl-fumarate in Multiple Sclerosis
Acronym: PRAG-MS
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: termination of the study due to the slowness of the recruitment activity, according to the contract signed with the Sponsor
Sponsor: Fondazione I.R.C.C.S. Istituto Neurologico Carlo Besta (Other)
Collaborators: Patient-Centered Outcomes Research Institute (Other); Universita degli Studi di Genova (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2017-000559-26
Record Dates: First submitted 2017-05-16; First posted 2017-11-17 (Actual); Last update posted 2019-10-31 (Actual); Status verified 2019-10

CONDITIONS: Relapsing Remitting Multiple Sclerosis
Keywords: Multiple Sclerosis
MeSH Terms: conditions — Multiple Sclerosis, Relapsing-Remitting; Multiple Sclerosis | interventions — Fingolimod Hydrochloride; Dimethyl Fumarate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Fingolimod 0.5 mg/day (Active Comparator): The study drugs, FTY and DMT, are approved and available on the market and safety and tolerability profile of both the drugs is well known. In our study, patients will be treated according to the clinical practice.
  Dose: FTY 0.5 mg/day or DMF 240 mg twice daily
  Interventions: Drug: Fingolimod
- Dimethyl Fumarate 240 mg twice daily (Active Comparator): The study drugs, FTY and DMT, are approved and available on the market and safety and tolerability profile of both the drugs is well known. In our study, patients will be treated according to the clinical practice.
  Dose: FTY 0.5 mg/day or DMF 240 mg twice daily
  Interventions: Drug: Dimethyl Fumarate

INTERVENTIONS:
Drug: Fingolimod — Fingolimod is a currently approved oral DMT for the treatment of relapsing remitting MS. It modulates sphingosine-1 phosphate receptors.
  Arms: Fingolimod 0.5 mg/day
Drug: Dimethyl Fumarate — Dimethyl Fumarate is a currently approved oral DMT for the treatment of relapsing remitting MS. The mode of action comprises immunomodulatory effects and an activation of nuclear (erythroid-derived 2) related factor mediated antioxidative response pathways leading to additional cytoprotective effects.
  Arms: Dimethyl Fumarate 240 mg twice daily

SUMMARY:
This will be a 1:1 randomized open label trial. European and outside Europe centres will be involved. Aim of the project is to conduct a head-to-head comparison of effectiveness of two approved disease modifying treatments (DMTs) in patients with relapsing remitting multiple sclerosis (RRMS). The term effectiveness refers to efficacy in a real life setting: this is intended to be in fact the first pragmatic multi-centre randomised controlled trial to directly assess the effectiveness of the new oral agents approved for MS (fingolimod/FTY versus dimethyl-fumarate/DMF) on disease activity, disability progression, quality of life, functioning and symptoms. It will be a randomized trial taking place in clinical care setting and comparing existing therapies, any of which may constitute standard care for naive patients or sub optimal responders to first-line drugs. Post hoc analysis will also identify the better treatment strategy on the different patient subgroups. Patient overall disease experience will be considered for the first time as the most important outcome. In fact, in addition to classical "no evidence of disease activity" (NEDA), a new composite NEDA taking account also of patient point of view and quality of life, will be proposed. Finally,the specific effectiveness profile of the two DMTs will be addressed, by exploring comparative benefits on different outcomes (disease activity, disability progression, brain atrophy, quality of life, fatigue, psychiatric and cognitive symptoms, medication satisfaction).

DETAILED DESCRIPTION:
Background and significance

1. The expansion of the treatment landscape in MS has increased the complexity of treatment decisions. Recommendations and algorithms can help to maximize the benefit of each available therapy; however, there is currently no consensus algorithm available, with most of the recently published recommendations being regional and most guidelines currently used in clinical practice, being driven by the labels of the therapies. The lack of head-to-head clinical trials for approved drugs is crucial since head-to-head trials constitute the gold standard for efficacy comparisons. This kind of information is mandatory for informed and objective health decisions. The present proposal aims at filling this critical gap in evidence. Randomized head-to-head trials are the best method for evaluating the efficacy of different treatments and to help the clinicians and the patients in health decision making. Randomized controlled trials, designed as experiments with high internal validity, have the ability to determine cause effect relationships. These experiments employ comprehensive designs to control for most, if not all, sources of bias by means of randomization, blinding, allocation concealment, etc. Usually, extended inclusion and exclusion criteria are used to identify a clearly defined population group of participants who would benefit from the intervention under investigation. Although the above experimental design, if correctly applied, leads to well-controlled trials with statistically credible results, the applicability of these results to real life practice may be questionable.

Here the investigators aim at conducting a comparative open label trial preserving the internal validity due to randomization and generalizability due to a pragmatic design. The term pragmatic is used for trials designed to test the effectiveness of the intervention in a broad routine clinical practice. The explanatory trial is designed in order to control for all known biases and confounders, so that the intervention's effect is maximized. The pragmatic trial, on the other hand, is designed to test interventions in the full spectrum of everyday clinical settings in order to maximize applicability and generalizability.1 This is intended to be the first pragmatic multi-centre randomised controlled trial to directly assess the effectiveness of the new oral agents approved for MS (FTY/gilenya versus DMF/tecfidera). FTY (0.5 mg/day) and DMF (240 mg twice daily) are both efficacious in the treatment of MS and both offer the convenience of an oral administration. As such they are similarly valuable alternative treatments for MS patients, and are indeed frequently proposed as possible alternative treatment options to MS patients. Indication for FTY is restricted in Europe to second line in first-line therapy non responders or in active naïve patients. DMF is highly prescribed also in active naive patients and as switching strategy in patients who do not adequately respond to self-injectable DMTs, such as FTY.

The need for randomized trials with approved drugs exists when treatment decision in clinical practice is challenged by the lack of evidence of superiority of one drug for a specific group of patients.

The efficacy profile of the two oral drug have been characterized in large clinical development programs. Oral therapies have been shown to offer benefits with regard to these clinical and MRI outcomes when compared with placebo in phase 3 trials.2-5 The clinical efficacy of these therapies over traditional injectable DMTs has been demonstrated for FTY in the trial assessing injectable interferon versus FTY720 oral in RRMS (TRANSFORMS).6 Findings of these phase 3 trials indicate that oral therapies may represent an advance in the treatment of MS because they offer effective treatment options that are often better tolerated and more convenient than the traditional injectable DMTs. There are no head-to-head controlled trials comparing the efficacy of the different oral DMTs. This is an area of much interest to neurologists and healthcare decision makers; therefore, indirect treatment comparisons have recently been performed. Of these, a recent study has compared FTY with DMF using a network meta-analysis approach and found no significant differences in relapse rate or in the proportion of patients with disability progression.7 Standard network meta-analysis methods may be susceptible to bias because of differences in trial populations and methodologies. Subgroup and post hoc analyses of the phase 3 trials of DMTs have demonstrated that differences in patient baseline characteristics influence the observed effect of DMTs on relapse rate and disability progression,6,8 and that the application of different definitions of disability progression has a large impact on disability outcomes.9 Therefore, it is important to adjust for these potentially confounding factors when assessing the comparative efficacy of these oral DMTs. It has been reported that FTY therapy results in a higher probability of no evidence of disease activity (NEDA) than DMF therapy when phase 3 trial data are indirectly compared and differences between trials are adjusted for.10 These findings must, however, be interpreted with caution, owing to the assumptions inherent in any modeling approach.

The need for high-quality, widely applicable evidence is gaining momentum, especially amidst health care policy makers. The increased costs of interventions and health care in a resource-limited environment have fueled the demand for clinically effective and applicable evidence. Here the investigators aim at conducting a comparative open label trial preserving the internal validity due to randomization and generalizability due to a pragmatic design. It will be the first randomized pragmatic trials in MS. Policy makers have an active interest in pragmatic trials, since these are designed to answer the question most relevant to a decision maker's agenda: comparative effectiveness of interventions in the routine practice. The availability of comparative data from routine practice will help policy makers to efficiently allocate resources and manpower and will drive patients and clinicians in shared and informed health decisions. The evolving MS landscape, in which a number of new treatments are appearing-each with their own benefits and risks-will require a change in the nature of interactions between patients and their physicians, with a shared approach to clinical decision making that emphasizes patient-related goals. Together, these innovations in MS management offer exciting new opportunities to optimize treatment outcomes. This will necessitate attention both to traditional clinical endpoints such as relapses and disability, to objective radiological surrogates of disease activity, and to newer outcome measures such as brain atrophy , cognition and patient-reported outcomes. In line with this, the present proposal aims at comparing the effectiveness of two oral MS agents on patient overall disease experience. If, traditionally, both clinical trials and routine medical care have relied on outcomes assessed by healthcare professionals, here the investigators want to focus also on the importance of self-evaluation of health, thus growing participation of individuals in their own care. The investigators can foresee a continuum where patient empowerment contributes to improve his/her healthcare and, at the same time, makes valuable medical data accessible to the medical community for future therapeutic developments.

The whole idea of applicable and generalizable research is very appealing and of benefit to the health sciences community.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with RRMS eligible to be treated with both FTY and DMF. Patients eligible for enrolment are patients for whom both drugs can be prescribed, upon clinical judgement and local label indication.
* Patients must be able to sign and date a written informed consent prior to entering the study. Where the subject is unable to write, consent may be given and recorded through appropriate alternative means in the presence of at least one impartial witness. In that case, the witness shall sign and date the informed consent document.
* Women of child-bearing potential must have a negative serum pregnancy test before enrollment and must practice an effective method of birth control, in line with normal clinical practice recommendations.

Exclusion Criteria:

* any FTY/DMF contraindication, as for authorized indications or clinical judgment;
* present immunodeficiency syndrome (primary or secondary immune deficiency);
* abnormal lymphocyte count;
* severe chronic active infections or acute infections not resolved at the time of the enrolment;
* evidence of active tuberculosis (TB);
* history of either untreated or inadequately treated latent TB infection;
* progressive Multifocal Leukoencephalopathy, even if only suspected;
* active malignancies;
* severe liver impairment (Child-Pugh class C);
* macular edema;
* sieronegative for antibodies IgG anti-VZV;
* hypersensitivity to the active substances or to any of the excipients;
* cardiac contraindications to FTY (patients who in the last 6 months experienced myocardial infarction, unstable angina, stroke, TIA, decompensated heart failure (HF) requiring hospitalization or Class III/IV HF; history or presence of Mobitz Type II second-degree or third-degree atrioventricular (AV) block or sick sinus syndrome, unless patient has a functioning pacemaker);
* pregnancy or breastfeeding;
* concomitant treatment with any other approved or investigational DMTs or other prohibited treatments.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 55 (Actual)
Dates: Start 2017-04-30 (Actual); Primary Completion 2019-10-30 (Actual); Study Completion 2019-10-30 (Actual)

PRIMARY OUTCOMES:
effectiveness of fingolimod 0.5 mg once daily versus dimethyl-fumarate 240 mg twice daily | 24 Months
  losing the NEDA status

SECONDARY OUTCOMES:
Annual relapse rate | over 12 and 24 months
  compare the effectiveness of the two oral DMTs in terms of prevention of clinical relapses
Number of Gd+ MRI lesions | at 12 and 24 months
  compare the effectiveness of the two oral DMTs in terms of prevention of MRI activity
Brain volume loss | at 12 and 24 months
  compare the effectiveness of the two oral DMTs in terms of prevention of brain atrophy
Prevention of sustained disability progression (EDSS worsening) | over 24 months
  percentage of patients with confirmed increase of 1 point on the EDSS scale
Prevention of Objective sustained disability progression | over 12 and 24 months
  percentage of patients with change in gait performance (limb range of motion) assessed by inertial sensors
Patient-NEDA | over 24 months
  Percentage of patients maintaining patient-NEDA status
Prevention of Cognitive decline | over 12 and 24 months
  Change in cognitive impairment index (CII) assessed by Brief Repeatable Battery of Neuropsychological tests (BRB-N)
Evaluation of social cognition | over 12 and 24 months
  Change in social cognition assessed by Story based Empathy task (SET)
Evaluation of quality of decision making | over 12 and 24 months
  Change in quality of decision making assessed by Game of Dice Task (GDT)
Preservation of Quality of life | over 12 and 24 months
  Multiple Sclerosis Quality of Life-54 (MSQOL-54) is a multidimensional health-related quality of life measure that combines both generic and MS-specific items into a single instrument. This 54-item instrument generates 12 subscales along with 2 summary scores, and 2 additional single-item measures. The MSQOL-54 is a structured, self-report questionnaire that the patient can generally complete with little or no assistance. MSQOL-54 scale scores are expressed on a 0-100 scale: higher scores indicating better functioning. There is no single overall score. Two summary scores, physical health and mental health, can be derived from a weighted combination of scale scores. In addition there are 12 subscales: physical function, role limitations-physical, role limitations-emotional, pain, emotional well-being, energy, health perceptions, social function, cognitive function, health distress, overall quality of life, sexual function and satisfaction with sexual function and change in health.
Convenience perception | over 12 and 24 months
  Convenience perception as measured by the convenience scale within Treatment Satisfaction Questionnaire for Medication-9 (TSQM-9). The scores in each domain of the TSQM-9 will be calculated as recommended by the instrument's authors (Atkinson MJ, et all. Health Qual Life Outcomes. 2004 Feb 26; 2:12)
Psychiatric symptoms | over 12 and 24 months
  Symptomatic changes as determinated by Hospital Anxiety & Depression Scale (HADS). HADS anxiety (HADS-A) and depression (HADS-D) scores range from 0 (no symptoms) to 21 (most severe Study Protocol, VS1 Page 26 of 48 symptoms).
Fatigue | over 12 and 24 months
  Symptomatic changes as determinated by Modified Fatigue Impact Scale (MFIS). The MFIS is a valid and reliable 21-question scale (score range, 0-84), with lower total scores indicating lower impact of fatigue on patient function.

CONTACTS AND LOCATIONS:
Overall Officials: Renato Mantegazza, MD, Principal Investigator — Fondazione IRCCS Istituto Neurologico Carlo Besta
Locations (1):
- Fondazione IRCCS Istituto Neurologico C. Besta, Neuroimmunology Unit, Milan, Italy

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Patsopoulos NA. A pragmatic view on pragmatic trials. Dialogues Clin Neurosci. 2011;13(2):217-24. doi: 10.31887/DCNS.2011.13.2/npatsopoulos. PMID 21842619
- [Background] Calabresi PA, Radue EW, Goodin D, Jeffery D, Rammohan KW, Reder AT, Vollmer T, Agius MA, Kappos L, Stites T, Li B, Cappiello L, von Rosenstiel P, Lublin FD. Safety and efficacy of fingolimod in patients with relapsing-remitting multiple sclerosis (FREEDOMS II): a double-blind, randomised, placebo-controlled, phase 3 trial. Lancet Neurol. 2014 Jun;13(6):545-56. doi: 10.1016/S1474-4422(14)70049-3. Epub 2014 Mar 28. PMID 24685276
- [Background] Kappos L, Radue EW, O'Connor P, Polman C, Hohlfeld R, Calabresi P, Selmaj K, Agoropoulou C, Leyk M, Zhang-Auberson L, Burtin P; FREEDOMS Study Group. A placebo-controlled trial of oral fingolimod in relapsing multiple sclerosis. N Engl J Med. 2010 Feb 4;362(5):387-401. doi: 10.1056/NEJMoa0909494. Epub 2010 Jan 20. PMID 20089952
- [Background] Fox RJ, Miller DH, Phillips JT, Hutchinson M, Havrdova E, Kita M, Yang M, Raghupathi K, Novas M, Sweetser MT, Viglietta V, Dawson KT; CONFIRM Study Investigators. Placebo-controlled phase 3 study of oral BG-12 or glatiramer in multiple sclerosis. N Engl J Med. 2012 Sep 20;367(12):1087-97. doi: 10.1056/NEJMoa1206328. PMID 22992072
- [Background] Gold R, Kappos L, Arnold DL, Bar-Or A, Giovannoni G, Selmaj K, Tornatore C, Sweetser MT, Yang M, Sheikh SI, Dawson KT; DEFINE Study Investigators. Placebo-controlled phase 3 study of oral BG-12 for relapsing multiple sclerosis. N Engl J Med. 2012 Sep 20;367(12):1098-107. doi: 10.1056/NEJMoa1114287. PMID 22992073
- [Background] Cohen JA, Barkhof F, Comi G, Hartung HP, Khatri BO, Montalban X, Pelletier J, Capra R, Gallo P, Izquierdo G, Tiel-Wilck K, de Vera A, Jin J, Stites T, Wu S, Aradhye S, Kappos L; TRANSFORMS Study Group. Oral fingolimod or intramuscular interferon for relapsing multiple sclerosis. N Engl J Med. 2010 Feb 4;362(5):402-15. doi: 10.1056/NEJMoa0907839. Epub 2010 Jan 20. PMID 20089954
- [Background] Hutchinson M, Fox RJ, Havrdova E, Kurukulasuriya NC, Sarda SP, Agarwal S, Siddiqui MK, Taneja A, Deniz B. Efficacy and safety of BG-12 (dimethyl fumarate) and other disease-modifying therapies for the treatment of relapsing-remitting multiple sclerosis: a systematic review and mixed treatment comparison. Curr Med Res Opin. 2014 Apr;30(4):613-27. doi: 10.1185/03007995.2013.863755. Epub 2013 Nov 26. PMID 24195574
- [Background] Giovannoni G, Cook S, Rammohan K, Rieckmann P, Sorensen PS, Vermersch P, Hamlett A, Viglietta V, Greenberg S; CLARITY study group. Sustained disease-activity-free status in patients with relapsing-remitting multiple sclerosis treated with cladribine tablets in the CLARITY study: a post-hoc and subgroup analysis. Lancet Neurol. 2011 Apr;10(4):329-37. doi: 10.1016/S1474-4422(11)70023-0. PMID 21397565
- [Background] Nixon R, Bergvall N, Tomic D, Sfikas N, Cutter G, Giovannoni G. No evidence of disease activity: indirect comparisons of oral therapies for the treatment of relapsing-remitting multiple sclerosis. Adv Ther. 2014 Nov;31(11):1134-54. doi: 10.1007/s12325-014-0167-z. Epub 2014 Nov 21. PMID 25414048
- See also: 9. Bergvall N, Sfikas N, Alsop J, Chin P, von Rosensteil P, Kappos L. Consequences of different definitions of confirmed disability progression across randomised trials of MS therapies. — http://novartis.medicalcongressposters.com/Default.aspx?doc=9ce32